CLINICAL TRIAL: NCT06646614
Title: Group Advanced Care Planning Pilot for Veterans
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Manali I. Patel, Staff Physician, VA Palo Alto Health Care System
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 67728
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The statistician analyzing the data will be masked from the experimental treatment and the control as will all research staff who are abstracting or collecting outcomes data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): The patient will continue to receive as normal and usual care. The participant will also receive educational materials in writing regarding advance care planning mailed to their preferred mailing address. The participants will complete surveys and interviews at baseline at again at 8 weeks post enrollment.
- Group Advance Care Planning (Experimental): The participant will engage in 2 hours of educational sessions regarding advance care planning and goals of care. They will be interviewed which is expected to last 20-30 min and surveys will last 15-20 min. The total involvement will be no more than 3 hours and 40 min over 8 weeks.
  Interventions: Behavioral: Group Advance Care Planning Education

INTERVENTIONS:
Behavioral: Group Advance Care Planning Education — Those assigned to the group ACP arm will receive usual care and the intervention which consists of 2 virtual or in-person sessions for a total of 2 hours by a trained community health worker/health educator. Sessions will introduce advanced care planning, help veterans discuss their goals of care with their care teams and learn how to discuss with their families and oncologist, and filing an advanced directive. Participants will be surveyed and interviewed at baseline and again at 8 months post-enrollment.
  Arms: Group Advance Care Planning

SUMMARY:
The proposed research aims to engage participants in group educational sessions to facilitate learning of topics related to advanced care planning and to determine whether this approach is more effective than usual care alone.

DETAILED DESCRIPTION:
The purpose of this study is to compare usual care against a group advanced care planning intervention comprised of two sessions led by trained community health workers or health educators from VA Palo Alto. A total of 60 participants will be randomly assigned to either usual care (n=30) or usual care + group advanced care planning intervention (n=30). Those in usual care will be mailed some educational materials about advanced care planning that they may review independently. Those in the group advanced care planning arm will participate in two 60-90 minute educational sessions led by a community health worker/educator that will either be conducted in person on-site, by VA-approved video conference, or a hybrid model. Topics will include an introduction to advanced care planning, goals of care topics, advance directives, and physicians order of life sustaining treatment. Both usual care and the group advanced care planning arms will also participate in pre/post surveys and/or interviews.

ELIGIBILITY:
Inclusion Criteria:

1. All patients >18 years old with newly diagnosed cancer are eligible.
2. Patients must have the ability to understand and willingness to provide verbal consent
3. Participants must speak English

Exclusion Criteria:

1. Inability to consent to the study
2. Plans to move within the area and leave the VA system within 4 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Goals of Care Documentation | Week 8 after patient enrollment
  Documentation of goals of care discussions will be analyzed for each patient at 8 weeks after patient enrollment.

SECONDARY OUTCOMES:
Feeling Heard and Understood | Baseline and Week 8 after patient enrollment
  Each patient will receive a validated Heard and Understood assessment survey. 4-item National Quality Forum-endorsed survey assessing self-perceived quality of communication with clinical care team. Each question is scored with a range of 0 to 4, with analyses comparing the proportion of patients reporting a top score (4) for a given question. The measure's reliability and validity has been assessed in a large study of outpatients with serious illness. It will be collected by self-report and self-administered assessment for each patient at Baseline and Week 8.
Change in patient activation using the Patient Activation Measure | Baseline and Week 8 after patient enrollment
  Each patient will receive a validated patient activation survey (PAM-13) to assess their activation. This is a validated measure from Insignia Health. Responses are: disagree strongly, disagree, agree, agree strongly with higher activation correlated with responses of agree and agree strongly. Each item is rated on 4-point scale (1 strongly disagree to 4 strongly agree, with additional "not applicable" option). Higher scores indicate greater patient activation. It will be collected for each patient by self-assessment at Baseline and Week 8.
Change in patient satisfaction with decision using the Satisfaction with Decision Measure | Baseline and Week 8 after patient enrollment
  Each patient will receive a validated satisfaction with decision survey to assess their satisfaction with decision. It will be analyzed for each patient at Baseline and Week 8.
Palliative Care Use (Self-reported and Chart Review) | At Baseline, 8 weeks and 6 months after patient enrollment
  Palliative care use will be analyzed for each patient at Week 8.
Hospice Care Use (Self-reported and Chart Review) | At Baseline, 8 weeks and 6 months after patient enrollment
  Hospice care use will be analyzed for each patient at Week 8.
Hospitalization Visits (Self-reported and Chart Review) | At Baseline, 8 weeks and 6 months after patient enrollment
  Hospital use for each patient will be self-reported by each patient or abstracted by electronic medical record at Week 8.

CONTACTS AND LOCATIONS:
Locations (1):
- VA Palo Alto, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No
We will not share.